CLINICAL TRIAL: NCT03556839
Title: A Randomized Phase III Trial of Platinum Chemotherapy Plus Paclitaxel With Bevacizumab and Atezolizumab Versus Platinum Chemotherapy Plus Paclitaxel and Bevacizumab in Metastatic (Stage IVB), Persistent, or Recurrent Carcinoma of the Cervix
Brief Title: Platinum Chemotherapy Plus Paclitaxel With Bevacizumab and Atezolizumab in Metastatic Carcinoma of the Cervix
Acronym: BEATcc
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other); Multicenter Italian Trials in Ovarian cancer and gynecologic malignancies (Unknown); MaNGO (Unknown); NSGO (Unknown); Japanese Gynecologic Oncology Group (Other); Gynecologic Oncology Group Foundation (Unknown); AGO Study Group (Other); Apices Soluciones S.L. (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-Cx10 / BEATcc; 2018-000367-83 (EudraCT Number); ENGOT-Cx10 (Other: ENGOT); GEICO 68-C (Other: GEICO); JGOG1084 (Other: JGOG); GOG-3030 (Other: GOG); 2024-514179-17-00 (EU CTIS Number)
Record Dates: First submitted 2018-05-18; First posted 2018-06-14 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma of the Cervix, Stage IVB
Keywords: Cervix; Carcinoma; Atezolizumab
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma | interventions — atezolizumab; Bevacizumab; Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Cisplatin 50mg/m2 or carboplatin AUC 5 + paclitaxel 175mg/m2+ bevacizumab 15mg/kg i.v D1 Q3W. Patients who achieve a complete response after ≥6 treatment cycles may be allowed to continue only on biologic therapy, namely bevacizumab, upon investigator discussion.
  Interventions: Drug: Bevacizumab; Drug: Cisplatin/Carboplatin; Drug: Paclitaxel
- Arm B (Experimental): cisplatin 50mg/m2 or carboplatin AUC 5 + paclitaxel 175mg/m2 + bevacizumab 15mg/kg + atezolizumab 1200mg i.v, D1 Q3W.Patients who achieve a complete response after ≥6 treatment cycles may be allowed to continue only on biologics therapy, namely bevacizumab plus atezolizumab, upon investigator discussion.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Cisplatin/Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Intravenous Infusion
  Other Names: Tecentriq
  Arms: Arm B
Drug: Bevacizumab — Intravenous Infusion
  Other Names: Avastin
Drug: Cisplatin/Carboplatin — Intravenous Infusion
Drug: Paclitaxel — Intravenous Infusion

SUMMARY:
The study will integrate the efficacy of combining the anti programmed death-ligand 1 (anti-PD-L1) agent atezolizumab with the current standard of care in Stage IVB , persistent or recurrent carcinoma of the cervix, namely cisplatin or carboplatin/paclitaxel/bevacizumab. It will be explored the combination of bevacizumab plus atezolizumab, with no patient selection based on PD-L1 expression, allowing an all-comer assessment of atezolizumab activity.

The study is a randomized open label phase III trial to investigate the impact of atezolizumab in combination with bevacizumab and cisplatin or carboplatin /paclitaxel chemotherapy on overall survival and will employ the intent to treat principle, and random assignment to one of the 2 arms will be balanced according to disease histology (squamous cell carcinoma vs adenocarcinoma), prior platinum therapy as a radiation sensitizer (no prior cis-Radiotherapy (RT) versus prior cis-RT) and chemotherapy backbone (cisplatin vs carboplatin).

This trial will be run in an open label design due to the following considerations: the control arm is the standard of care for women diagnosed with metastatic, persistant or recurrent cervical cancer because of its impact on overall survival and the primary endpoint of the study is overall survival (OS), so blinding is not needed to ensure a robust assessment.

DETAILED DESCRIPTION:
Given that both Vascular Endothelial Growth Factor (VEGF) and PD-L1 appear important in cervical cancer pathogenesis, this study is designed to test the hypothesis that breaking of immune tolerance by PD-1/PD-L1 blockade will enhance the efficacy of anti-VEGF therapy in the treatment of patients with metastatic , persistent or recurrent cervical cancer. There are several data suggesting that atezolizumab and bevacizumab may be synergistic. Enhanced tumor angiogenesis is commonly associated with absence of tumor-infiltrating T cells in patients. There is evidence in ovarian cancer that tumor expression of VEGF is negatively correlated to the density of CD8+ TILs and this phenotype is associated with early recurrence, consistent with prior studies showing a correlation of VEGF to early recurrence and short survival. Furthermore, in ascites, high levels of VEGF correlate to low numbers of NK T-like CD3+CD56+ cells.

In addition to promoting tumor angiogenesis, there is increasing evidence that VEGF plays a role in cancer immune evasion through several different mechanisms. Indeed, emerging evidence suggests that the endothelium acts as a selective barrier, allowing certain T cell subsets, notably T regulatory (Treg) cells, to traffic more effectively into the tumor contributing to tumor immune tolerance. In addition, some experiments have shown that tumour hypoxia promotes the recruitment of regulatory T (T reg) cells through induction of expression of the chemokine CC-chemokine ligand 28 (CCL28), which, in turn, promotes tumour tolerance and angiogenesis.

Some immunosuppressive activities of VEGF, however, can be reversed by inhibition of VEGF signaling. Mice exposed to pathophysiologic levels of VEGF exhibited impaired dendritic cell function, which could be restored by blockade of VEGFR2.

In turn, the anti-tumor effect of angiogenesis blockade requires CD8+ T cells supporting the notion that VEGF-A do not simply promote tumor growth through angiogenesis. Thus, peripheral immune tolerance and angiogenesis programs seem closely connected and cooperating to sustain tumour growth.

In addition, there is evidence that anti-VEGF therapy and immunotherapy act synergistically. Motz et al have suggested that the combination of anti-VEGF-A antibody and immunotherapy with adoptive T cell transfer led to a superior infiltration of tumor-reactive T cells than any single approach. Indeed, in a murine melanoma model, VEGF blockade synergized with adoptive immunotherapy, as evidenced by improved anti-tumor activity, prolonged survival, and increased trafficking of T cells into tumors. These data are reminiscent of the additive benefit observed in patients by combining recombinant interferon-alpha therapy and bevacizumab, a recombinant, humanized therapeutic antibody directed against VEGF, for the treatment of metastatic renal cell carcinoma.

More evidence has come from a clinical study of subjects with melanoma combining the checkpoint inhibitor (anti-CTLA-4) ipilimumab and bevacizumab. In 46 patients, the combined therapy yielded a 19.6% objective response rate, stable disease in 13%. All responses were durable >6 months and median survival was 25.1 months, much prolonged compared to ipilimumab's expectation in metastatic melanoma. Activated vessel endothelium with extensive CD8+ T cell and macrophage cell infiltration was observed in post-treatment biopsies, as well as marked increases in CD4/CCR7/CD45ROm central memory cells in peripheral blood in the majority of patients.

Thus, an emerging paradigm supported by the data above is that angiogenesis and immune suppression are two facets of a linked biological program. Tumors seem to co-opt these existing mechanisms that are normally required to limit excessive inflammation and promote tissue recovery during infection or wound healing. The execution of this program sustains tumor growth and promotes immunologic tolerance. Because of the intimate relationship between angiogenesis and immunosuppression, it is thus expected that inhibiting both pathways will result in improved and more durable clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients must be ≥18 years of age.
2. Signed informed consent before any study-specific procedure
3. Able (in the investigator´s judgment) to comply with the study protocol
4. GOG/Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. Life expectancy ≥3 months
6. Histologically- or cytologically-confirmed diagnosis of metastatic (stage IVB), persistent, or recurrent cervical cancer (histologies other than squamous cell, adenocarcinoma, or adenosquamous will be excluded) not amenable for curative treatment with surgery and/or radiation therapy. The inclusion of patients with adenocarcinoma histology will be capped to 20% of the whole study population.
7. No prior systemic anti-cancer therapy for metastatic or recurrent disease.
8. Measureable disease by RECIST v1.1 criteria.
9. A tumor specimen is mandatory at study entry.
10. Adequate organ function:

    Hemoglobin ≥9 g/dL ANC ≥1.5 × 109/L Lymphocyte count ≥0.5 × 109/L Platelet count ≥100 x 109/L
11. Adequate liver function:

    Serum albumin ≥2.5 g/dL Total serum bilirubin ≤1.5 ×ULN AST and ALT ≤2.5 × upper limit normal (ULN) or ≤5 × ULN if tumor involvement (liver) is present
12. Adequate renal function:

    Patients with serum creatinine <1.5 × ULN Urine dipstick for proteinuria <2+.
13. Adequate coagulation:

    Blood coagulation parameters (PTT, PT/INR): PT such that international normalized ratio (INR) is ≤ 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thromboembolus) and a PTT <1.5 × ULN.
14. Negative Test Results for Hepatitis:

    Negative hepatitis B surface antigen (HBsAg) test at screening Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening.The HBV DNA test will be performed only for patients who have a positive total HBcAb test.

    Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening.The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
15. Toxicities related to previous treatments must be recovered to < grade 2 (with the exception of alopecia).
16. Female participants must be postmenopausal (≥ 12 months of non-therapy-induced amenorrhoea) or surgically sterile (absence of ovaries and/or uterus, or who received therapeutic radiation to the pelvis) or otherwise have a negative serum pregnancy test within 7 days of the first study treatment and agree to abstain from heterosexual intercourse or use single or combined contraceptive methods that result in a failure rate of <1% per year during the whole treatment period of the study and for at least 5 months (if the last study dose contained atezolizumab) or 6 months (if the last study dose contained bevacizumab) after the last dose of study treatment.

    * Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal or postovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

1. Disease that is suitable for local therapy administered with curative intent
2. Prior radiotherapy delivered using cobalt (rather than a linear accelerator)
3. Patients with Stage IVA not amendable to concurrent chemo-radiation as primary treatment will not be eligible.
4. Ongoing disease involving the bladder or rectum at screening/baseline
5. Evidence of abdominal free air
6. Bilateral hydronephrosis, unless it can be alleviated by ureteral stent(s) or percutaneous drainage
7. Patients previously treated with chemotherapy except when used concurrently with radiation therapy. Patients who have received either concurrent paclitaxel with radiation therapy or carboplatin/paclitaxel as adjuvant therapy are ineligible for the study.
8. Prior treatment with any anti-VEGF drug, including bevacizumab, CD137 agonists or immune checkpoint blockade therapies, anti-PD1, or anti-PDL1 therapeutic antibodies or anti-CTLA 4.
9. Patients with a concomitant malignancy other than non-melanoma skin cancer. Patients with a prior invasive malignancy (except non-melanoma skin cancer ) who have had any evidence of disease within the last 5 years or whose prior malignancy treatment contraindicates the current protocol therapy.
10. Known brain metastases or spinal cord compression. It is mandatory to perform a scan of the brain in cases of suspected brain metastases (CT or MRI) or spinal cord compression (MRI).
11. History or evidence, following a neurological examination, of central nervous system (CNS) disorders, unless properly treated with standard medical treatment,(e.g. uncontrolled epileptic seizures). History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study.
12. Patients with serious non-healing wound, ulcer, or bone fracture.
13. Acute intestinal obstruction or sub-occlusion episode in the last 6 months.
14. Active GI bleeding or GI ulcer
15. History of Crohn's disease or inflammatory bowel disease
16. Prior bowel resection ≤6 weeks preceding first study dose
17. History of diverticulitis requiring medical intervention
18. NCI CTCAE (version 5.0) grade ≥2 enteritis
19. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1, Cycle 1.
20. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1, Cycle 1.
21. Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
22. Current or recent (within 10 days before the first dose of study drug) chronic daily treatment with aspirin (>325 mg/day), clopidogrel (>75 mg/day), or current or recent (within 10 days before first dose of bevacizumab) use of therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes.
23. Patients with pre-existing Grade 2 or greater peripheral neuropathy.
24. History of any grade ≥3 venous thromboembolic event (VTE)
25. Patients with clinically significant cardiovascular disease.
26. Left ventricular ejection fraction defined by MUGA/ECHO below the institutional lower limit of normal.
27. Uncontrolled tumor-related pain
28. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
29. Uncontrolled hypercalcemia (>1.5 mmol/L ionized calcium or calcium >12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.
30. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, glomerulonephritis or celiac disease.

    History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
31. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
32. Active tuberculosis
33. Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
34. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
35. Received therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1
36. Known human immunodeficiency virus (HIV)
37. Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study Influenza vaccination should be given during influenza season only
38. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
39. Treatment with systemic immunostimulatory agents (including but not limited to IFNs, IL-2) within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1
40. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1 The use of corticosteroids is allowed as premedication for paclitaxel-based regimen. All patients should be premedicated prior to receiving chemotherapy (including with corticosteroids) according to the prescription information of paclitaxel and cisplatin/carboplatin and the institutional standard of care guidance.
41. Currently participating or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of study treatment.
42. Prior anti-cancer monoclonal antibody (mAb), prior chemotherapy, targeted small molecule therapy as first line treatment for the treatment of metastatic or recurrent cervical cancer.
43. Women that are breastfeeding or pregnant
44. Known hypersensitivity to bevacizumab, atezolizumab or any of theirs excipients (including Cremophor)
45. Demonstration of any other neurological or metabolic dysfunction, found upon physical examination or laboratory tests involving a reasonable suspicion of the existence of a disease or condition that contraindicates the use of an experimental drug, or that involves an increased risk to the patient of treatment-related complications
46. No medical or psychiatric illness that may impede the performance of a systemic or surgical treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 410 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 48 months
  Time from the date of randomization to the date of first documentation of disease progression or death due to any cause, whichever occurs first based on investigator assessment using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1)
Overall survival | 48 months
  Time from the date of randomization to the date of death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate | 48 months
  Based on investigator assessment using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1)
Duration of response | 48 months
  Based on investigator assessment using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1)
Incidence of Treatment-Emergent Adverse Events of combining atezolizumab to chemotherapy plus bevacizumab compared to cisplatin or carboplatin/paclitaxel (CP) plus bevacizumab. | 48 months
  Incidence, nature and severity of adverse events (AEs) assessed by CTCAE version 5.0
First subsequent therapy | 48 months
  Time from randomization to first subsequent therapy or death due to any cause
Progression-free survival 2 | 48 months
  Time from randomization to the second event of disease progression per radiological criteria, start of a new line of therapy, due to symptomatic deterioration or to death due to any cause
Patient-reported outcomes (PROs) of function and health related quality of life (HR-QOL) associated with atezolizumab + CP + bevacizumab compared to bevacizumab + CP alone, as measured by the functional and GHS/ HRQoL scales of EORTC QLQ-C30 | 48 months
  Mean and mean changes from baseline score in patient function (role, physical) and GHS/HRQoL, by assessment timepoint and between treatment arms, as assessed by the functional and GHS/HRQoL scales of EORTC QLQ-C30.
Pharmacokinetics (PK) of atezolizumab | 36 months
  Serum concentration (Cmin) of atezolizumab
Pharmacokinetics (PK) of atezolizumab | 36 months
  Serum concentration (Cmax) of atezolizumab
Incidence of anti-therapeutic antibodies (ATAs) | 36 months
  Incidence of ATAs during the study relative to the prevalence of ATAs at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ana Oaknin, MD PhD, Principal Investigator — Vall d´Hebron University Hospital
Locations (72):
- United States (2):
  - Willis Knighton Cancer Center, Shreveport, Louisiana
  - Massey Cancer Center, Richmond, Virginia
- France (17):
  - ICO Paul Papin, Angers
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Hôpital Privé du Confluent S.A.S., Nantes
  - Centre Antoine Lacassagne, Nice
  - Groupe Hospitalier Diaconesses-Croix Saint-Simon, Paris
  - HEGP, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO-HPCA, Plérin
  - ICO Centre René Gauducheau, Saint-Herblain
  - Hôpitaux Universitaires, Strasbourg
  - Institut Claudius Régaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (2):
  - Universitätsmedizin Mainz, Mainz
  - Helios-Klinikum Wuppertal, Wuppertal
- Italy (17):
  - Fondazione Del Piemonte Per L'Oncologia, Candiolo
  - Azienda Ospedaliero-Universitaria Di Ferrara, Ferrara
  - Ospedale Lecce 'Vito Fazzi', Lecce
  - ASST Lecco, Lecco
  - Irst Irccs, Meldola FC
  - Irccs S. Raffaele - Milano, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Gerardo, Monza
  - Istituto Nazionale Tumori Di Napoli Irccs Pascale, Napoli
  - Istituto Oncologico Veneto (IOV) IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - AUSL Romagna - P.O. di Ravenna, Lugo, Faenza, Rimini e Cattolica, Ravenna
  - Azienda Usl - Irccs Di Reggio Emilia, Reggio Emilia
  - Policlinico Universitario A. Gemelli, Roma
  - AOU Città della Salute e della Scienza di Torino, Presidio Sant'Anna, Torino
  - Ospedale Ordine Mauriziano, Torino
  - Azienda Sanitaria Universitaria Integrata Di Udine, Udine
- Japan (8):
  - Kurume University Hospital, Fukuoka
  - Saitama medical university international medical center, Hidaka
  - Hokkaido Cancer Center, Hokkaido
  - Hyogo Cancer Center, Hyōgo
  - Cancer Institute Hospital, Kōtoku
  - Niigata University Medical & Dental Hospital, Niigata
  - Shizuoka Cancer Center, Shizuoka
  - Keio University Hospital, Tokyo
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
- Spain (19):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Intitut Català d' Oncolgia L' Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Donostia- Donostia Unibertsitate Ospitalea, Donostia / San Sebastian, Gipuzkoa
  - Hospital de la Vall d'Hebron, Barcelona
  - H. Clínic Barcelona, Barcelona
  - Hospital Reina Sofía Cordoba, Córdoba
  - ICO Girona, Girona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Regional de Málaga, Málaga
  - Hospital Clinico Universitario Virgen Arrixaca, Murcia
  - Hosptial Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Quirón de Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza
- Sweden (4):
  - Lindköping University Hospital, Linköping
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takekuma M, Nishio S, Yamaguchi S, Yunokawa M, Nishio H, Nishino K, Kurosaki A, Minobe S, Villacampa G, Oaknin A, Okamoto A. Atezolizumab, bevacizumab, and platinum chemotherapy in cervical cancer: results of Japanese population from BEATcc. J Gynecol Oncol. 2025 Nov;36(6):e116. doi: 10.3802/jgo.2025.36.e116. Epub 2025 May 19. PMID 40968753
- [Derived] Oaknin A, Gladieff L, Martinez-Garcia J, Villacampa G, Takekuma M, De Giorgi U, Lindemann K, Woelber L, Colombo N, Duska L, Leary A, Godoy-Ortiz A, Nishio S, Angelergues A, Rubio MJ, Farinas-Madrid L, Yamaguchi S, Lorusso D, Ray-Coquard I, Manso L, Joly F, Alarcon J, Follana P, Romero I, Lebreton C, Perez-Fidalgo JA, Yunokawa M, Dahlstrand H, D'Hondt V, Randall LM; ENGOT-Cx10-GEICO 68-C-JGOG1084-GOG-3030 Investigators. Atezolizumab plus bevacizumab and chemotherapy for metastatic, persistent, or recurrent cervical cancer (BEATcc): a randomised, open-label, phase 3 trial. Lancet. 2024 Jan 6;403(10421):31-43. doi: 10.1016/S0140-6736(23)02405-4. Epub 2023 Dec 1. PMID 38048793
- [Derived] Grau JF, Farinas-Madrid L, Oaknin A. A randomized phase III trial of platinum chemotherapy plus paclitaxel with bevacizumab and atezolizumab versus platinum chemotherapy plus paclitaxel and bevacizumab in metastatic (stage IVB), persistent, or recurrent carcinoma of the cervix: the BEATcc study (ENGOT-Cx10/GEICO 68-C/JGOG1084/GOG-3030). Int J Gynecol Cancer. 2020 Jan;30(1):139-143. doi: 10.1136/ijgc-2019-000880. Epub 2019 Oct 23. PMID 31645423